CLINICAL TRIAL: NCT02033187
Title: Phase 4 Study of the Impact of Daily Bathing With Chlorhexidine-gluconate Impregnated Bathing Cloths on Nosocomial Infections in Critically Ill Patients
Brief Title: Daily Chlorhexidine Bathing and Infection Rates in Critically-ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Michael Noto, Clinical Fellow, Division of Allergy, Pulmonary, and Critical Care Medicine, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 120502
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Healthcare Associated Infections
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorhexidine bathing (Experimental): Patients in an ICU randomized to treatment arm 1 will be bathed with single use, no rinse, disposable cloths impregnated with 2% chlorhexidine gluconate solution (Sage® 2% Chlorhexidine Gluconate Cloths). Bathing of the skin of the arms, chest, abdomen, back, both legs, perineum, and buttocks will be performed daily and as needed after patients become soiled. The face and neck will not be bathed in this manner but will be bathed with water-moistened washcloths. All other infection control and cleaning procedures will be performed per the current practice in each intensive care unit.
  Interventions: Other: Chlorhexidine bathing
- Non-chlorhexidine bathing (Active Comparator): Patients in an ICU randomized to treatment arm 2 will be bathed with single use, no rinse, disposable cloths that do not contain chlorhexidine gluconate solution (Sage Comfort Bath® Cleansing Washcloths). Bathing of the skin of the arms, chest, abdomen, back, both legs, perineum, and buttocks will be performed daily and as needed after patients become soiled. The face and neck will not be bathed in this manner but will be bathed with water-moistened washcloths. All other infection control and cleaning procedures will be performed per the current protocols in each intensive care unit.
  Interventions: Other: Non-chlorhexidine bathing

INTERVENTIONS:
Other: Chlorhexidine bathing — Patients in an ICU randomized to treatment arm 1 will be bathed with single use, no rinse, disposable cloths impregnated with 2% chlorhexidine gluconate solution (Sage® 2% Chlorhexidine Gluconate Cloths). Bathing of the skin of the arms, chest, abdomen, back, both legs, perineum, and buttocks will be performed daily and as needed after patients become soiled. The face and neck will not be bathed in this manner but will be bathed with water-moistened washcloths. All other infection control and cleaning procedures will be performed per the current practice in each intensive care unit.
  Arms: Chlorhexidine bathing
Other: Non-chlorhexidine bathing — Patients in an ICU randomized to treatment arm 2 will be bathed with single use, no rinse, disposable cloths that do not contain chlorhexidine gluconate solution (Sage Comfort Bath® Cleansing Washcloths). Bathing of the skin of the arms, chest, abdomen, back, both legs, perineum, and buttocks will be performed daily and as needed after patients become soiled. The face and neck will not be bathed in this manner but will be bathed with water-moistened washcloths. All other infection control and cleaning procedures will be performed per the current protocols in each intensive care unit.
  Arms: Non-chlorhexidine bathing

SUMMARY:
Healthcare-associated infections are a major cause of morbidity among critically ill patients. Bathing critically ill patients with cloths impregnated with the broad-spectrum antimicrobial agent chlorhexidine-gluconate may decrease healthcare-associated infections. The purpose of this study is to evaluate the effect of daily bathing with disposable chlorhexidine-impregnated bathing cloths, as compared to daily bathing with disposable standard non-chlorhexidine-impregnated bathing cloths, on the rates of healthcare-associated infections in critically-ill patients.

Hypothesis: Daily bathing of the skin with chlorhexidine-impregnated bathing cloths will result in reduced rates of healthcare-associated infections in patients admitted to intensive care units (ICU).

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the medical, surgical, trauma, cardiovascular and neuro adult intensive care units at Vanderbilt University Medical Center

Exclusion Criteria:

1. Being cared for in the burn ICU or patients with TEN/SJS or burns being cared for in one of the non-burn intensive care units.
2. Patients with known allergy to chlorhexidine gluconate
3. Age < 18 years old
4. Patients where daily bathing would not be safe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12000 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
A composite of healthcare-associated infections | Daily
  A composite of the following healthcare-associated infections:
  1. Central line-associated blood stream infections (CLABSI)
  2. Possible or probable ventilator associated pneumonia (VAP)
  3. Catheter-associated urinary tract infection (CAUTI)
  4. C. difficile-associated diarrhea

SECONDARY OUTCOMES:
Rates of each individual site infection included in the composite calculation above | Daily
  1. Central line-associated blood stream infections (CLABSI)
  2. Possible or probable ventilator associated pneumonia (VAP)
  3. Catheter-associated urinary tract infection (CAUTI)
  4. C. difficile-associated diarrhea
Skin reactions | As needed
  Skin reactions related to topical chlorhexidine
Hospital mortality | One year
  Hospital mortality
Hospital length of stay | One year
  Hospital length of stay
ICU length of stay | One year
  ICU length of stay
Rate of cultures positive for multi-drug resistant organisms | Daily
Rates of blood culture contamination | Daily
Rates of healthcare-acquired bloodstream infections | Daily

OTHER OUTCOMES:
Subgroup analysis by the individual intensive care unit | One year

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Noto, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Noto MJ, Domenico HJ, Byrne DW, Talbot T, Rice TW, Bernard GR, Wheeler AP. Chlorhexidine bathing and health care-associated infections: a randomized clinical trial. JAMA. 2015 Jan 27;313(4):369-78. doi: 10.1001/jama.2014.18400. PMID 25602496